CLINICAL TRIAL: NCT01068444
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase II Study to Assess the Efficacy and Safety of Pioglitazone in Patients With Nonalcoholic Steatohepatitis
Brief Title: The Efficacy and Safety of Pioglitazone in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Long Chuang, M.D., Ph D., Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUH-HB9608
Record Dates: First submitted 2010-02-11; First posted 2010-02-15 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis
Keywords: NASH; Pioglitazone; Treatment
MeSH Terms: conditions — Hepatitis | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental): Pioglitazone 30 mg/day for 6 months and 3 months of follow-up period after treatment
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Placebo 30 mg/day for 6 months and 3 months of follow-up period after treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pioglitazone — 1. Name: GLITOS（Pioglitazone）
  2. Dosage form: Tablets
  3. Dose(s): 30mg
  4. Dosing schedule: QD
  5. Duration: 6 months
  Other Names: GLITOS
  Arms: Pioglitazone
Drug: placebo — placebo 30 mg/d for 6 months
  Arms: Placebo

SUMMARY:
Recent studies have demonstrated that PPARγ as well as diet control could improve glycemic control, decrease serum ALT level, decrease hepatic fat distribution, and increase intrahepatic insulin sensitivity. The purposes of this study are:

1. Primary aims:

1. Comparison between Pioglitazone and placebo groups in terms of steatosis and liver function tests.
2. Evaluation of clinical safety of Pioglitazone

2. Secondary aims:

1. Comparison between Pioglitazone and placebo groups in terms of liver necroinflammation and fibrosis.
2. The impact of Pioglitazone on the related metabolic index, including insulin resistance(HOMA-IR), newly-onset diabetes, metabolic syndrome, lipid profiles (T-Chol, HDL-C, LDL-C, TG).
3. Comparison between Pioglitazone and placebo groups in terms of high-sensitive C-reactive protein changes.

3. Interventional aim: Assessment the association between magnetic resonance imaging study and intrahepatic fat distribution before and after Pioglitazone treatment.

DETAILED DESCRIPTION:
Pioglitazone belongs to thiazolidinediones and anti-diabetes drug which decreases the insulin resistance. It increases the use of glucose of peripheral tissues and decrease the production of glucose from liver and dose not influence the production of insulin. It is agonist of peroxisome proliferator-activated receptor-gamma (PPARγ) and by binding to the receptors of PPARγ in various tissues it has effects on transcription of the insulin-dependent gene. In animal model, pioglitazone has shown to influence the metabolism by the insulin-dependent mechanism.

Recent studies have demonstrated that PPARγ as well as diet control could improve glycemic control, decrease serum ALT level, decrease hepatic fat distribution, and increase intrahepatic insulin sensitivity. Meanwhile, PPARγ could also prevent the development of alcohol-induced steatohepatitis, improve hepatic necroinflammatory activity, and decrease lipid deposition. It is not yet clearly known how the effect of P-PARγ agonist among Asian peoples.

ELIGIBILITY:
Main inclusion criteria:

1. Male and female patients with 18-70 years of age
2. Liver biopsy findings consistent with the diagnosis of NASH with or without compensated cirrhosis within one year before baseline
3. Compensated liver disease
4. Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
5. All fertile males and females must be using two forms of effective contraception during treatment during the 3 months after treatment.
6. ALT level between 1.3-5 x ULN for 2 occasions during 6 months before screening.
7. HbA1C ≦ 8.0 during screening

Main exclusion criteria:

1. Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) *6 months before baseline.
2. History or other evidence of a medical condition associated with chronic liver disease other than NASH (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, > 20 g/day for female or > 40 g/day for male, toxin exposures)
3. hepatocellular carcinoma
4. History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
5. Serum creatinine level >1.5 times the upper limit of normal at screening and calculated creatinine clearance as calculated by Cockcroft and Gault < 60mL/min during screening
6. History of ischemic heart disease during screening
7. New York Heart Association (NYHA) Functional Class 1-4 cardiac status during screening
8. Albumin <3.2g/dL during screening
9. Total bilirubin >1.2 x ULN during screening. Patients with history of asymptomatic indirect hyperbilirubinemia whose total bilirubin < 2 x ULN and direct bilirubin < 20% of total bilirubin could be included.
10. History of prothrombin time > 15 seconds or International normalized ratio (INR) > 1.3
11. Organ, stem cell, or bone marrow transplant
12. History of serious concurrent medical illness that in the investigator's opinion might interfere with therapy this includes significant systemic illnesses (other than liver disease) such as chronic pancreatitis
13. Active systemic autoimmune disorder
14. Pregnancy (or lactation) or, in subjects capable of bearing children, inability / unwillingness to practice adequate contraception
15. Females of child-bearing potential (post-puberty) unwilling or unable to have pregnancy testing at any study visit
16. Therapy with a systemic antiviral agent (with the exception of prophylaxis or treatment of influenza or chronic HSV) within the past 30 days prior to screening.
17. Concurrent participation in another clinical trial in which the subject is or will be exposed to another investigational or a non-investigational drug or device within 6 weeks of the screening visit
18. Current therapy with insulin within 1 week prior to screening.
19. Experienced use with PPARg agonist (e.g., rosiglitazone, pioglitazone) within 6 months prior to screening.
20. Known hypersensitivity to any component of PPARg agonists
21. A history of hepatotoxicity to TZDs and/or a history of severe edema or a medically serious fluid-related event associated with the use of TZDs
22. History of metformin use within 3 months prior to screening.
23. Type Ⅰ diabetes
24. Seropositive of HBsAg, anti-HCV or anti-HIV during screening or 3 month prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-04; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Comparison between Pioglitazone and placebo groups in terms of steatosis and liver function tests | 9 months
Evaluation of clinical safety of Pioglitazone | 9 months

SECONDARY OUTCOMES:
Comparison between Pioglitazone and placebo groups in terms of liver necroinflammation and fibrosis. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Long Chuang, MD, PhD, Principal Investigator — Kaohsiung Medical University
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Municipal Hsiao-Kang Hospital, Kaohsiung Medical University, Kaohsiung City

REFERENCES:
- [Derived] Huang JF, Dai CY, Huang CF, Tsai PC, Yeh ML, Hsu PY, Huang SF, Bair MJ, Hou NJ, Huang CI, Liang PC, Lin YH, Wang CW, Hsieh MY, Chen SC, Lin ZY, Yu ML, Chuang WL. First-in-Asian double-blind randomized trial to assess the efficacy and safety of insulin sensitizer in nonalcoholic steatohepatitis patients. Hepatol Int. 2021 Oct;15(5):1136-1147. doi: 10.1007/s12072-021-10242-2. Epub 2021 Aug 12. PMID 34386935
- [Derived] Huang JF, Yeh ML, Huang CF, Huang CI, Tsai PC, Tai CM, Yang HL, Dai CY, Hsieh MH, Chen SC, Yu ML, Chuang WL. Cytokeratin-18 and uric acid predicts disease severity in Taiwanese nonalcoholic steatohepatitis patients. PLoS One. 2017 May 4;12(5):e0174394. doi: 10.1371/journal.pone.0174394. eCollection 2017. PMID 28472039